CLINICAL TRIAL: NCT04790786
Title: The UPMC OPtimizing Treatment and Impact of Monocolonal antIbodieS Through Evaluation for COVID-19 Trial
Brief Title: UPMC OPTIMISE-C19 Trial, a COVID-19 Study
Acronym: OPTIMISE-C19
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Emergency Use Authorizations for monoclonal antibodies withdrawn
Sponsor: Erin McCreary (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Erin McCreary, Clinical Assistant Professor, University of Pittsburgh Medical Center
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY21020179
Record Dates: First submitted 2021-02-26; First posted 2021-03-10 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Covid19
Keywords: COVID; monoclonal antibodies
MeSH Terms: conditions — COVID-19 | interventions — imdevimab; etesevimab; sotrovimab; bebtelovimab

STUDY DESIGN:
Intervention Model Description: The study is an adaptive platform and as such is intended to study multiple interventions simultaneously, does not have a defined sample size, and is intended to move forward in perpetual fashion with domains and interventions being added and subtracted over time. For example, interventions will be added and subtracted depending on federal decisions regarding monoclonal antibodies, such as granting or revoking authorization for use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Lilly Bamlanivimab (Experimental): The Lilly monoclonal antibody bamlanivimab will be administered according to FDA EUA guidelines. Dosing is 700 mg intravenously times one within 10 days of COVID-19 symptom onset.
  Interventions: Biological: Lilly Bamlanivimab
- Regeneron Casirivimab + Imdevimab (Experimental): The Regeneron monoclonal antibody cocktail Casirivimab + Imdevimab will be administered according to FDA EUA guidelines. Dosing is 1200 mg of each drug (2400 mg total) administered intravenously times one within 10 days of COVID-19 symptom onset.
  Interventions: Biological: Regeneron Casirivimab + Imdevimab
- Lilly Bamlanivimab + Etesevimab (Experimental): The Lilly monoclonal antibody cocktail of bamlanivimab + etesevimab will be administered according to FDA EUA guidelines. Dosing is given intravenously times one within 10 days of COVID-19 symptom onset.
  Interventions: Biological: Lilly Bamlanivimab + Etesevimab
- Sotrovimab (Experimental): The monoclonal antibody of sotrovimab will be administered according to FDA EUA guidelines. Dosing is given intravenously times one within 7 days of COVID-19 symptom onset.
  Interventions: Biological: Sotrovimab
- Bebtelovimab (Experimental): The monoclonal antibody of bebtelovimab will be administered according to FDA EUA guidelines. Dosing is given intravenously times one within 7 days of COVID-19 symptom onset.
  Interventions: Biological: Bebtelovimab

INTERVENTIONS:
Biological: Lilly Bamlanivimab — Administration of Lilly Bamlanivimab to COVID positive patients
  Arms: Lilly Bamlanivimab
Biological: Regeneron Casirivimab + Imdevimab — Administration of Regeneron Casirivimab + Imdevimab to COVID positive patients
  Arms: Regeneron Casirivimab + Imdevimab
Biological: Lilly Bamlanivimab + Etesevimab — Administration of Lilly Bamlanivimab + Etesevimab to COVID positive patients
  Arms: Lilly Bamlanivimab + Etesevimab
Biological: Sotrovimab — Administration of Sotrovimab to COVID positive patients
  Arms: Sotrovimab
Biological: Bebtelovimab — Administration of Bebtelovimab to COVID positive patients
  Arms: Bebtelovimab

SUMMARY:
Multiple monoclonal antibodies (mABs) have been shown to reduce viral burden and improve clinical outcomes, have been granted FDA Emergency Use Authorization (EUA) for use in select populations, and are routinely used in the UPMC Health System, which has made expanded access a priority. However, the comparative effectiveness of these mABS is unknown. The National Academies of Sciences, Engineering, and Medicine has called for expanded access and clinical use of mABs, noting it is "critical to collect data and evaluate whether they are working as predicted". This pragmatic evaluation will determine the relative effects of the EUA-governed mABs versus each other. When U.S. government mAB policies change (e.g., FDA grants or revokes EUAs), UPMC Health System policies and the evaluated mABs will accordingly change.

DETAILED DESCRIPTION:
While COVID-19 vaccination will reduce COVID-19-related morbidity and mortality, the learned immune response may vary between individuals. This means interventions such as monoclonal antibodies (mAB) will still be needed to prevent progression of COVID-19 illness. Monoclonal antibodies seek to mimic or enhance the natural immune system response against a pathogen and are often used in the care of patients with cancer or infection.

For viral infections, mABs are created by exposing a white blood cell to a particular viral protein, which is then cloned to mass produce antibodies to target that virus. For SARS-CoV-2, the virus that causes COVID-19, IgG1 mABs target the spike protein of SARS-CoV-2 and block viral attachment and entry into cells.

The SARS-CoV-2 mABs bamlanivimab and etesevimab, and the REGN-COV2 combination (casirivimab + imdevimab) reduce nasopharyngeal viral burden plus clinical outcomes including future emergency department visits and hospitalizations. Each received FDA Emergency Use Authorization (EUA) for use in selected populations.

As of February 2021, there are over 60,000 new cases of COVID-19 diagnosed daily in the US, with over 7000 daily COVID-19 related hospital admissions. Although case volumes are currently declining, COVID-19 remains a significant public health threat.

Despite the EUAs, the clinical use of mABs is low due in part to lack of patient access, complexities in drug allocation, and lack of knowledge among providers are contributing factors. Further, the comparative effectiveness of different mABs is unknown and not yet directly studied. The National Academies of Sciences, Engineering, and Medicine recently called for expanded access and clinical use of mABs, noting it is "critical to collect data and evaluate whether they are working as predicted". This evaluation seeks to determine their relative effects versus each other, starting with those governed by EUAs.

OPTIMISE-C19 is a quality improvement (QI) study, governed by approvals from both the UPMC QI committee and the University of Pittsburgh IRB. Currently, mAB therapy is approved for use under EUA issued by the FDA. There are no data on the relative benefits of one mAB versus any other. mABs are ordered by UPMC physicians as a generic referral order and the order is filled by UPMC pharmacy via therapeutic interchange. The selection of mABs available within pharmacy is overseen by the UPMC pharmacy and therapeutics committee. OPTIMISE-C19 provides the therapeutic interchange via random allocation. The UPMC Quality Improvement Committee approved the OPTIMISE-C19 study, including the random therapeutic interchange. The University of Pittsburgh IRB considered the randomized therapeutic interchange to be quality improvement and approved the additional data collection and analyses.

Patients provide verbal consent to receive mAB therapy. UPMC requires physicians to provide and review with patients the EUA Fact Sheet for each mAB, and explain that the patient could receive any of the EUA-governed mABs. As per EUA requirements, physicians discuss the risks and benefits of mABs with patients, and patients consent to receive a mAB as part of routine care, should they desire mAB treatment. Patients are told which mAB they are receiving, and physicians and patients can agree to the assigned mAB or request a specific mAB. It is the treating physicians' and patients' choice to accept the assigned mAB or not. The QI committee considered these steps to represent adequate consent to participate. The IRB considered that the provision of mAB therapy therefore fell under quality improvement and only the additional data collection and analyses represented research. The IRB waived any additional consent requirements.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients
* Eligible for mAB under FDA EUA

Exclusion Criteria:

* Death is deemed to be imminent or inevitable
* Previous participation in this REMAP within the last 90 days

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4571 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCreary, PharmD, Study Director — University of Pittsburgh; David T Huang, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data underlying the results reported in journal articles, subject to appropriate security controls, may be available for sharing with other researchers.
Supporting Information: SAP
Time Frame: Relevant data may be available 1 year following publication
Access Criteria: Data access is subject to a methodologically sound proposal and the necessary data sharing agreements.

REFERENCES:
- [Derived] Huang DT, McCreary EK, Bariola JR, Minnier TE, Wadas RJ, Shovel JA, Albin D, Marroquin OC, Kip KE, Collins K, Schmidhofer M, Wisniewski MK, Nace DA, Sullivan C, Axe M, Meyers R, Weissman A, Garrard W, Peck-Palmer OM, Wells A, Bart RD, Yang A, Berry LR, Berry S, Crawford AM, McGlothlin A, Khadem T, Linstrum K, Montgomery SK, Ricketts D, Kennedy JN, Pidro CJ, Nakayama A, Zapf RL, Kip PL, Haidar G, Snyder GM, McVerry BJ, Yealy DM, Angus DC, Seymour CW. Effectiveness of Casirivimab-Imdevimab and Sotrovimab During a SARS-CoV-2 Delta Variant Surge: A Cohort Study and Randomized Comparative Effectiveness Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220957. doi: 10.1001/jamanetworkopen.2022.20957. PMID 35834252
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] McCreary EK, Bariola JR, Minnier TE, Wadas RJ, Shovel JA, Albin D, Marroquin OC, Kip KE, Collins K, Schmidhofer M, Wisniewski MK, Nace DA, Sullivan C, Axe M, Meyers R, Weissman A, Garrard W, Peck-Palmer OM, Wells A, Bart RD, Yang A, Berry LR, Berry S, Crawford AM, McGlothlin A, Khadem T, Linstrum K, Montgomery SK, Ricketts D, Kennedy JN, Pidro CJ, Haidar G, Snyder GM, McVerry BJ, Yealy DM, Angus DC, Nakayama A, Zapf RL, Kip PL, Seymour CW, Huang DT. The comparative effectiveness of COVID-19 monoclonal antibodies: A learning health system randomized clinical trial. Contemp Clin Trials. 2022 Aug;119:106822. doi: 10.1016/j.cct.2022.106822. Epub 2022 Jun 11. PMID 35697146
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Huang DT, McCreary EK, Bariola JR, Wadas RJ, Kip KE, Marroquin OC, Koscumb S, Collins K, Shovel JA, Schmidhofer M, Wisniewski MK, Sullivan C, Yealy DM, Axe M, Nace DA, Haidar G, Khadem T, Linstrum K, Snyder GM, Seymour CW, Montgomery SK, McVerry BJ, Berry L, Berry S, Meyers R, Weissman A, Peck-Palmer OM, Wells A, Bart R, Albin DL, Minnier T, Angus DC. The UPMC OPTIMISE-C19 (OPtimizing Treatment and Impact of Monoclonal antIbodieS through Evaluation for COVID-19) trial: a structured summary of a study protocol for an open-label, pragmatic, comparative effectiveness platform trial with response-adaptive randomization. Trials. 2021 May 25;22(1):363. doi: 10.1186/s13063-021-05316-3. PMID 34034784

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Started | 128 | 2454 | 885 | 1104
Completed | 128 | 2454 | 885 | 1104
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab | Total
Number analyzed (Participants) | 128 | 2454 | 885 | 1104 | 4571
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (17) | 54 (18) | 56 (16) | 53 (18) | 54 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 1320 | 470 | 599 | 2458
  Male | 59 | 1134 | 415 | 505 | 2113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 252 | 148 | 161 | 576
  White | 104 | 2089 | 693 | 892 | 3778
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 113 | 44 | 51 | 217

OUTCOME MEASURES:

1. Primary Outcome: Hospital-free Days
Description: Days alive and free from hospitalization. Patients that are both living and not in the hospital will meet criteria to be counted in this outcome. Deaths were rare and therefore the upper and lower end of the IQR are both 28, in addition to the median. This outcome measure does reflect median hospital free days and interquartile ranges for all groups.
Time Frame: 28 days after initial participation
Population: Every patient who received mAb treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 128 | 2454 | 885 | 1104
days | 28 [28 to 28] | 28 [28 to 28] | 28 [28 to 28] | 28 [28 to 28]
Statistical Analysis 1: Comparison: Lilly Bamlanivimab vs Regeneron Casirivimab + Imdevimab vs Lilly Bamlanivimab + Etesevimab vs Sotrovimab; The primary analysis model was a Bayesian cumulative logistic model that adjusted for treatment location (infusion center or ED), age (<30, 30-39, 40-49, 50-59, 60-69, 70-79, and ≥ 80 years), sex, and time (2-week epochs). Comparisons between individual mAb were based on the relative odds ratio between a given two arms for the primary outcome. An odds ratio for an arm to a comparator >1 implies improved outcomes. A sliding scale with different levels of equivalence bounds was pre-defined; Test type: Equivalence — Equivalence between two arms was defined as 95% posterior probability the odds ratio is within a given bound; Bayesian cumulative logistic model — Equivalence between two arms was defined as 95% posterior probability the odds ratio is within a given bound based on Bayesian probability; Bayesian cumulative logistic model, Equivalence between two arms was defined as 95% posterior probability the odds ratio is within a given bound; Equivalence between two arms was defined as 95% posterior probability the odds ratio is within a given bound

2. Secondary Outcome: All-cause Mortality at 28 Days
Description: All-cause mortality at 28 days.
Time Frame: 28 days after initial participation
Measure: Count of Participants; unit: Participants
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 128 | 2454 | 885 | 1104
Participants | 1 | 12 | 7 | 7

3. Secondary Outcome: SARS-CoV-2 Nasopharyngeal Viral Loads
Description: Where feasible SARS-CoV-2 nasopharyngeal viral loads among participants from baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab | Bebtelovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: SARS-CoV-2 Plasma Viral Loads
Description: Where feasible SARS-CoV-2 plasma viral loads among participants from baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab | Bebtelovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: SARS-CoV-2 Antibody Titers
Description: Where feasible SARS-CoV-2 antibody titers at baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: SARS-CoV-2 Antibody Neutralization
Description: Where feasible SARS-CoV-2 antibody neutralization at baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: SARS-CoV-2 Immune Responses
Description: Where feasible SARS-CoV-2 immune responses at baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Detection of SARS-CoV-2 Variants Through Next-generation Sequencing
Description: Where feasible detection of SARS-CoV-2 variants through next-generation sequencing at baseline and longitudinally through day 28
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Duration of SAR-CoV-2 Infectivity
Description: Where feasible determining the duration of SAR-CoV-2 infectivity among patients with persistent nasopharyngeal swab viral shedding
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Non-culture Surrogates for SARS-CoV-2 Infectivity
Description: Where feasible determining non-culture surrogates for SARS-CoV-2 infectivity among patients with persistent nasopharyngeal swab viral shedding
Time Frame: 28 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Non-culture Surrogates for SARS-CoV-2 Infectivity
Description: as for outcome 10
Time Frame: 90 days after initial participation
Population: Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Duration of SAR-CoV-2 Infectivity
Description: as for outcome 9
Time Frame: 90 days after initial participation
Population: Analysis not feasible due to limitations of pandemic, Participants were not consented for samples due to limited trial resources, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: ED Visit Within 28 Days
Time Frame: Duration of study
Population: Not feasible due to nature of data and treatment sites during pandemic, data not collected
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were reported by treating clinicians at each treatment center in a secure, nonpunative, system safety database and adjudicated by study researchers
Arm/Group | Lilly Bamlanivimab | Regeneron Casirivimab + Imdevimab | Lilly Bamlanivimab + Etesevimab | Sotrovimab
All-Cause Mortality (participants affected / at risk) | 1/128 | 12/2454 | 7/885 | 7/1104
Serious Adverse Events (participants affected / at risk) | 0/128 | 7/2454 | 0/885 | 4/1104
Other Adverse Events (participants affected / at risk) | 0/128 | 17/2454 | 12/885 | 6/1104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lilly Bamlanivimab (N=128) | Regeneron Casirivimab + Imdevimab (N=2454) | Lilly Bamlanivimab + Etesevimab (N=885) | Sotrovimab (N=1104)
chest pain (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) — chest pain during infusion reaction
other infusion reaction (Product Issues) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lilly Bamlanivimab (N=128) | Regeneron Casirivimab + Imdevimab (N=2454) | Lilly Bamlanivimab + Etesevimab (N=885) | Sotrovimab (N=1104)
infusion reaction (Product Issues) | 0 (0) | 17 (17) | 12 (12) | 6 (6)

LIMITATIONS AND CAVEATS:
Results are presented before any prespecified statistical trigger was reached. Lack of patient-level variant data limited ability to assess comparative effectiveness relative to variant strains. The EHR eligibility screen identified most, but not all, EUA risk factors and could not identify if a patient was asymptomatic or severely ill. Finally, vaccination status was unable to be ascertained for this cohort which may impact effectiveness of monoclonal antibody therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Bam-etes vs bam (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT04790786/Prot_SAP_001.pdf
  • Statistical Analysis Plan: cas-imd (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04790786/SAP_002.pdf